CLINICAL TRIAL: NCT02640170
Title: Intraoperative Imaging With ICG Registry
Status: Completed | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: UPCC 16915
Record Dates: First submitted 2015-12-22; First posted 2015-12-28 (Estimated); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Lung Nodule, Breast, Kidney,Parathyroid, Mediastinal, Skin Mass, Soft Tissue, Prostate, Stomach Pleural, Head and Neck, and Are at Risk of Recurrence
MeSH Terms: interventions — Registries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Registry

SUMMARY:
The purpose of this registry is to monitor the rate of recurrence in patients who undergo cancer surgery.

DETAILED DESCRIPTION:
Our objective is to collect prospective data on cancer subjects who undergo surgery and intraoperative imaging. The registry will include (but not limited to) cancer type, stage, intraoperative challenges to the surgeon, usage and results of intraoperative imaging, and recurrence surveillance.

In this protocol, subjects that receive intraoperative imaging will provide us the opportunity to record what tissues fluoresce in the operating room, and then to identify if these lesions are cancer when the histopathology is performed. Also, we will monitor any side effects or potential toxicities that may occur. This data can then be used to predict if a subject is more likely to develop a local recurrence due to missed cancer cells, metastatic lymph nodes or synchronous lesions.

ELIGIBILITY:
Inclusion Criteria:

Inclkusion Criteria

* Adult patients >= 18 years of age
* Patients presenting with any solid tumor and/or diseased tissue even benign nodules presumed to be resectable and are at risk for recurrence.
* Good operative candidate as determined by the treating physician and/or multidisciplinary team
* Subject capable of giving informed consent and participating in the process of consent.

Exclusion Criteria None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of any resectable solid tumor, including but not limited to lung nodule, breast, kidney,parathyroid, mediastinal, skin mass, soft tissue, prostate, stomach pleural, head and neck, and are at risk of recurrence
Sampling Method: Probability Sample
Enrollment: 291 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2020-02 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
Number of subjects registered | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Sunil Singhal, MD, PhD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Newton AD, Predina JD, Corbett CJ, Frenzel-Sulyok LG, Xia L, Petersson EJ, Tsourkas A, Nie S, Delikatny EJ, Singhal S. Optimization of Second Window Indocyanine Green for Intraoperative Near-Infrared Imaging of Thoracic Malignancy. J Am Coll Surg. 2019 Feb;228(2):188-197. doi: 10.1016/j.jamcollsurg.2018.11.003. Epub 2018 Nov 22. PMID 30471345